CLINICAL TRIAL: NCT03746327
Title: English Efficacy and Tolerance of 4 Weeks of Tedizolid in Prosthetic Joint Infections Treated With Implant Removal
Brief Title: Efficacy and Tolerance of 4 Weeks of Tedizolid in Prosthetic Joint Infections Treated With Implant Removal
Acronym: PROTEDI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Anna Cruceta, Project manager, Fundacion Clinic per a la Recerca Biomédica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROTEDI 2018-002465-18
Record Dates: First submitted 2018-07-26; First posted 2018-11-19 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-03

CONDITIONS: Prostheses Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sivextro arm (Experimental): 200 mg milligram per day during 4 weeks
  Interventions: Drug: Sivextro 200 milligrams Oral Tablet

INTERVENTIONS:
Drug: Sivextro 200 milligrams Oral Tablet — 200 mg milligram per day during 4 weeks

SUMMARY:
To evaluate the efficacy of 4 weeks of 200 mg/24h of tedizolid for prosthetic join infections caused by tedizolid susceptible microorganisms treated with implant removal in one or two stages at 6 months of followup after stopping tedizolid treatment.

DETAILED DESCRIPTION:
To evaluate the efficacy of 4 weeks of 200 mg/24h of tedizolid for prosthetic join infections caused by tedizolid susceptible microorganisms treated with implant removal in one or two stages at 6 months of followup after stopping tedizolid treatment.

Secondary objectives:

Evaluate the efficacy of tedizolid at 12 months of follow-up; evaluate the rate of gastrointestinal adverse events with tedizolid; determine the rate of haematological abnormalities during tedizolid treatment and; in case of two-stage exchange, the rate of positive cultures during reimplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female older than 18 years who accept and sign the informed consent.
2. Infection signs onset more than 3 months after index arthroplasty.
3. Diagnostic of chronic (≥3 weeks of clinical symptoms) hip or knee prosthetic joint infection according to MSIS criteria *(Parvizi J, Gherke T. Definition of peri-prosthetic joint infection. J Arthroplasty 2014; 29: 1331)
4. Infection due to a tedizolid susceptible microorganism.
5. Surgical approach: one or two - stage exchange of all implant components.
6. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Patients with a prosthetic joint infection with negative cultures.
2. Patients who undergo debridement without removing the prosthesis or only partially removed
3. ≥15 days of other antibiotic treatment before starting tedizolid
4. Life expeancy ≤ 1 year.
5. Previous enrollment in this protocol.
6. Hypersensitivity to tedizolid or any formulation excipients.
7. Concurrent use of another investigational medication within 30 days of study entry.
8. Women who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Investigator-assessed incidence of local signs infection at 6 months after tedizolid | 6 months
  incidence or absence of local signs of infection at the 6 months after tedizolid treatment.

SECONDARY OUTCOMES:
Incidence of Adverse Events at 12 months after ending tedizolid treatment | 12 months
  incidence of adverse events at the 12 months after tedizolid treatment. number of Adverse Events as assessed
Incidence of positive blood cultures during reimplantation on the two stage exchange cases. | 0, 7 days and months 1, 2, 6, 12
  incidence blood cultures at reimplantation,

CONTACTS AND LOCATIONS:
Locations (1):
- Laura Morata, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided